CLINICAL TRIAL: NCT04383925
Title: Randomized Trial Evaluating the Non-specific Effects of Different BCG Strains in Guinea-Bissau: Effects on Early-life Mortality and Morbidity
Brief Title: Trial to Compare Two Strains of BCG
Acronym: STRAIN III
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BCGSTRAIN III; 071/CNES/INASA/2020 (Registry Identifier: The Nacional Committee for Ethics in Health of Guinea-Bissau); 2002944 (Registry Identifier: The Developing-Country Committee of The National Committee on Health Research Ethics in Denmark)
Record Dates: First submitted 2020-05-04; First posted 2020-05-12 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Death, Infant; Morbidity;Infant
Keywords: BCG vaccination; Non-specific effects of BCG; Heterologous effects; Maternal immune priming
MeSH Terms: conditions — Infant Death

STUDY DESIGN:
Intervention Model Description: Outcome assessor-blinded RCT
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Following informed consent, the mother selects, from a stack of envelopes, a closed envelope that contains a sealed randomization lot indicating allocation to either BCG-Japan or BCG-Russia. The mother, inclusion assistant and vaccinator will thus not be blinded to the intervention allocation. All assistants assessing outcomes during the follow-up procedures outlined and providers of care will be blinded to the randomization allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCG-Japan (Experimental): Infants randomized to receive BCG-Japan at discharge from the Maternity Ward will receive one 0.05 ml dose of Mycobacterium bovis BCG live attenuated vaccine BCG-Japan (Tokyo BCG Laboratory) by intradermal injection in the left deltoid region. Dependent on national supply, infants will receive oral polio vaccine (OPV) at the time of BCG vaccination.
  Interventions: Biological: BCG-Japan
- BCG-Russia (Active Comparator): Infants randomized to receive BCG-Russia at discharge from the Maternity Ward will receive one 0.05 ml dose Mycobacterium bovis BCG live attenuated vaccine BCG-Russia-I (Serum Institute of India) by intradermal injection in the left deltoid region. Dependent on national supply, infants will receive oral polio vaccine (OPV) at the time of BCG-vaccination.
  Interventions: Biological: BCG-Russia

INTERVENTIONS:
Biological: BCG-Japan — Infant (<1 year) 0.05 ml dose of resuspended BCG-Japan (Tokyo strain 172, Japan BCG Laboratory, 1-5-21 Otsuka, Bunkyo-ku, Tokyo, 112-0012 Japan).
  Other Names: Tokyo strain 172
  Arms: BCG-Japan
Biological: BCG-Russia — Infant (<1 year) 0.05 ml dose of resuspended BCG-Russia (Serum Institute of India)
  Arms: BCG-Russia

SUMMARY:
The trial will be a two-year outcome assessor-blinded RCT at the maternity ward of hospital Simão Mendes (HNSM) in urban Bissau, Guinea-Bissau to compare BCG-Japan versus BCG-Russia 1:1 in 15,000 infants with respect to mortality, morbidity and case-fatality rate during hospital admission. The trial will also examine the association between BCG strains and BCG skin reaction characteristics by six weeks (data collected by telephone) and at two and six months (data collected at home-visits to a subgroup of the cohort).

As a secondary aim, this large study will be used to further evaluate the role of maternal BCG immune priming for overall health, since there are indications that maternal BCG scarring enhances the non-specific effects of BCG.

DETAILED DESCRIPTION:
This two-year outcome assessor-blinded RCT will be conducted at the maternity ward of hospital Simão Mendes (HNSM) in urban Bissau, Guinea-Bissau to compare BCG-Japan versus BCG-Russia 1:1 in 15,000 infants with respect to mortality, morbidity and case-fatality rate during hospital admission.

The trial will also examine the association between BCG strains and BCG skin reaction characteristics by six weeks (data collected by telephone) and at two and six months (data collected at home-visits to a subgroup of the cohort).

HYPOTHESES

The aim is to investigate the following hypotheses:

1. Compared with BCG-Russia, receiving BCG-Japan is associated with

   1. a 16% reduction in all-cause deaths and
   2. a 10% lower case-fatality rate for hospitalized infants.
2. BCG-vaccinated children have lower mortality if the mother has a BCG scar, when compared to if the mother does not have a BCG scar.

METHODS Setting: The RCT will be carried out by the Bandim Health Project (BHP) in a close collaboration with the HNSM Maternity Ward. BHP maintains a Health and Demographic Surveillance System (HDSS) site in Guinea-Bissau, covering approx. 100,000 individuals in six suburbs of the capital Bissau. A dedicated BHP team registers all births and vaccinations at the Maternity Ward, where BHP has conducted a series of RCTs since 2002, with the aim of improving early-life health outcomes.

Inclusion: Neonates born at the HNSM Maternity Ward and neonates referred to the ward for vaccination are eligible for participation in the study.

Mothers/guardians to infants eligible for the study will receive an oral study explanation in Portuguese Creole and a written explanation in Portuguese. Provided that oral consent is obtained, the mother/guardian signs a written consent form; if the mother or guardian is illiterate, a fingerprint can be provided to confirm participation. The family can request that their child leaves the trial at any time. Infants that are not eligible for participation or whose mother/guardian declines participation will be registered and vaccinated by our team (standard practice). Information on maternal and paternal BCG scar status, scar size, mid-upper-arm circumference and socioeconomic factors will be collected during the inclusion procedure.

Telephone contact information for the mother, the father and family members and/or persons living in the same house are recorded at inclusion. BCG will be provided at discharge for all infants at the ward.

Randomization:

Following informed consent, the mother selects, from a stack of envelopes, a closed envelope that contains a sealed randomization lot indicating allocation to either BCG-Japan or BCG-Russia. The mother, inclusion assistant and vaccinator will thus not be blinded to the intervention allocation.

Vaccination: The infant is vaccinated intradermally with 0.05 ml of the allocated BCG strain in the left upper deltoid, followed by vaccination with OPV. OPV is provided via the National Vaccination Program; if OPV is in shortage, only BCG vaccination will be provided.

Follow-up:

All assistants assessing outcomes during the follow-up procedures outlined below will be blinded to the randomization allocation.

Follow-up takes place through three mechanisms:

1. All enrolled infants with a telephone number recorded at inclusion: Family telephone interview at 6 weeks and 6 months to register dates and outcomes of consultations, hospital admissions and whether the child died. If the child died, the mother/guardian is briefly asked about symptoms and whether the death occurred at home or at a hospital. Information on adherence to the 6-week vaccination schedule, infant BCG reaction status and adverse events is also collected. If the infant has not yet received the 6-week vaccines, the mother/guardian will be reminded that it is time for the infant to be vaccinated.
2. Cohort of BHP HDSS infants: home visits at 2 and 6 months of age. With the proposed sample size of 15,000 infants and an estimated 15.5% residing in the HDSS study area, the trial will enroll approximately 2,300 children from the HDSS. These children will be followed by our routine surveillance system and receive two additional home visits at 2- and 6 months of age. At the visits, data is collected on mortality, morbidity, BCG scar status and size, adverse events and maternal and paternal BCG scar status (if not collected at inclusion).
3. All enrolled infants: Registration of admissions and consultations at the HNSM pediatric ward.

Admissions, diagnoses and outcomes at the pediatric ward are documented by a BHP team on all days of the year. Parental names and telephone numbers are registered for all admissions.

Sample size:

Primary outcome: Based on BCGSTRAIN I trial data and BCGSTRAIN II trial data (unpublished), an overall mortality rate of 1.1% by 6 weeks of age is anticipated. Given that two large-scale RCTs testing BCG-Japan vs. BCG-Russia have been conducted in Guinea-Bissau, the sample size needed to demonstrate a significant difference in all-cause mortality between BCG-Japan and BCG-Russia has been calculated based on the conditional power of a meta-analysis involving BCGSTRAIN I, II and a third RCT, as detailed by Roloff et al. In order to detect a 16% reduction in all-cause mortality associated with BCG-Japan in the meta-analysis of the three RCTs, with an expected heterogeneity of 0.002 between the trials, a conditional power of 0.80 and an alpha of 0.05, an additional 148 events in the third trial is necessary. With an expected mortality rate of 1.1%, this corresponds to a sample size of 15,000 inclusions when considering an expected loss to follow-up of approx. 10%.

With an expected monthly inclusion rate of 600 infants based on previous experiences, it is expected that at least 15,000 children, i.e. 7,500 in each BCG strain group, can be included during an expected timeframe of approx. 2 years for inclusion procedures and an additional 6 months for follow-up procedures.

Analyses:

The mortality and morbidity data will be analyzed as intention-to-treat in Cox regression models with age as the underlying time variable. In-hospital case-fatality rates between BCG strains will be compared using Fischer's exact test (2-sided). In case an OPV or vitamin A supplementation campaign or similar campaigns with potential immune stimulatory effects occurs during the study period, the main comparison of the two strains and of the effects of maternal BCG scarring on infant outcomes will be conducted by censoring all children on the first day of the campaign, to exclude any interaction of the campaign with the BCG strains.

As sensitivity analyses, an analysis where same-day deaths and admissions (events occurring on the day of BCG vaccination) are omitted will be conducted. An analysis of main outcomes excluding neonates that were admitted to intensive care before inclusion will also be conducted.

All analyses will be conducted overall and stratified by maternal BCG scar status and sex.

Trial vaccines:

The BCG vaccines will be acquired from the Japan BCG laboratory (BCG-Japan) and the Serum Institute of India (BCG-Russia).

Ethical considerations:

The proposed study will randomize children to BCG strains that are distributed by UNICEF and widely used in Guinea-Bissau and the rest of the world. Our previous studies have shown that providing BCG vaccination at discharge is safe and beneficial. Oral and written informed consent will be obtained in all cases. The study protocol was approved by the Ethical Committee in Guinea-Bissau and the Central Ethical Committee in Denmark gave its consultative approval. A local clinical monitor will be appointed to oversee the study.

Public health importance:

Global annual infant BCG vaccinations exceed 120 million. Current BCG vaccine strains are heterogeneous due to accumulation of genetic diversity and non-standardized production techniques. Yet, there is a substantial lack of data comparing the various BCG strains both in terms of specific and non-specific effects.

By providing information regarding BCG strains and data on the importance of maternal immune priming with BCG, the proposed study is likely to be an important contribution to future BCG policies. Substantial improvements in protection from TB and reductions in early-life morbidity and mortality will likely be achieved at low cost, if more information on the efficacy of the different strains of BCG and the importance of maternal immune priming is made available.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants present at the HNSM maternity ward on the day of discharge or procuring vaccination at the ward.

Exclusion Criteria:

* Infants older than 6 weeks (>42 days) of age
* Infants that have already received either BCG or oral polio vaccine (OPV)
* Infants that are moribund due to gross malformation or acute illness (about to die or be transferred to the pediatric ward according to the local health physician assessment; the latter children may be recruited when they are discharged from the pediatric ward or the neonatal intensive care unit).

Ages: 0 Days to 42 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16390 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Rate of all-cause mortality overall and stratified by maternal BCG scar status and sex | Six weeks of age
  Data on mortality is collected from all available information sources (admission at HNSM, telephone follow-up, HDSS data)

SECONDARY OUTCOMES:
Rate of hospital admissions overall and stratified by maternal BCG scar status and sex | Six weeks and six months of age
  Data on hospital admissions is collected at HNSM's Pediatric Ward
In-hospital case-fatality risk ratio overall and stratified by maternal BCG scar status and sex | Six weeks and six months of age
  Data on hospital admission and in-hospital case-fatality among admitted infants is collected at HNSM's Pediatric Ward
Prevalence of BCG skin reactions | Six weeks and six months of age
  The effect of the BCG strains on the BCG skin reaction prevalence will be evaluated by six weeks and six months of age. The data is obtained from telephone follow-up.
Prevalence of BCG skin reactions | Six weeks and six months of age
  The effect of the BCG strains on the BCG skin reaction prevalence by two months and six months of age. The data is obtained from home visits to infants residing in the BHP HDSS.
Prevalence of different BCG skin reaction types | Two and six months of age
  The effect of the BCG strains on the BCG skin reaction type. The reaction types are papules, pustules, scars and no reaction. Data is obtained from home visits to infants residing in the BHP HDSS.
Size of BCG skin reactions | Two and six months of age
  The effect of the BCG strains on the BCG skin reaction size. Data is obtained from home visits to infants residing in the BHP HDSS.
Rate of adverse events | 6 months
  To register adverse events from BCG vaccination in the form of simple or suppurative lymphadenitis, mothers are given a detailed explanation of these conditions and they are encouraged at inclusion and at subsequent follow-up visits to bring their child to a HDSS health center for consultation if such a condition should arise. Furthermore, mothers are asked at the time of telephone follow-up whether their child has or had a swollen lymph node in the left armpit and if yes, whether there has been secretion. At HDSS study area home visits, mothers are equally asked, and the size of the axillary lymph node is examined. A size <16 mm will be considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, Professor, Principal Investigator — Bandim Health Project; Christine Stabell Benn, Professor, Study Chair — Bandim Health Project, University of Southern Denmark; Frederik Schaltz-Buchholzer, MD, Study Director — Bandim Health Project, University of Southern Denmark
Locations (1):
- Bandim Health Project, Bissau, Guinea-Bissau

IPD SHARING:
Plan to Share IPD: Yes
The trial steering committee can share individual participant data after after approval of a data sharing agreement sent to cbenn@health.sdu.dk
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year after follow-up procedures have been completed.
Access Criteria: The trial steering committee can be approached for data sharing at cbenn@health.sdu.dk

REFERENCES:
- [Background] Wardlaw T, You D, Newby H, Anthony D, Chopra M. Child survival: a message of hope but a call for renewed commitment in UNICEF report. Reprod Health. 2013 Dec 11;10:64. doi: 10.1186/1742-4755-10-64. PMID 24325885
- [Background] Lawn JE, Cousens S, Zupan J; Lancet Neonatal Survival Steering Team. 4 million neonatal deaths: when? Where? Why? Lancet. 2005 Mar 5-11;365(9462):891-900. doi: 10.1016/S0140-6736(05)71048-5. PMID 15752534
- [Background] Calmette A. Preventive Vaccination Against Tuberculosis with BCG. Proc R Soc Med. 1931 Sep;24(11):1481-90. doi: 10.1177/003591573102401109. No abstract available. PMID 19988326
- [Background] Benn CS, Roth A, Garly ML, Fisker AB, Schaltz-Buchholzer F, Timmermann A, Berendsen M, Aaby P. BCG scarring and improved child survival: a combined analysis of studies of BCG scarring. J Intern Med. 2020 Dec;288(6):614-624. doi: 10.1111/joim.13084. Epub 2020 May 25. PMID 32301189
- [Background] Roth A, Sodemann M, Jensen H, Poulsen A, Gustafson P, Weise C, Gomes J, Djana Q, Jakobsen M, Garly ML, Rodrigues A, Aaby P. Tuberculin reaction, BCG scar, and lower female mortality. Epidemiology. 2006 Sep;17(5):562-8. doi: 10.1097/01.ede.0000231546.14749.ab. PMID 16878042
- [Background] Timmermann CA, Biering-Sorensen S, Aaby P, Fisker AB, Monteiro I, Rodrigues A, Benn CS, Ravn H. Tuberculin reaction and BCG scar: association with infant mortality. Trop Med Int Health. 2015 Dec;20(12):1733-44. doi: 10.1111/tmi.12614. Epub 2015 Oct 22. PMID 26426863
- [Background] Garly ML, Martins CL, Bale C, Balde MA, Hedegaard KL, Gustafson P, Lisse IM, Whittle HC, Aaby P. BCG scar and positive tuberculin reaction associated with reduced child mortality in West Africa. A non-specific beneficial effect of BCG? Vaccine. 2003 Jun 20;21(21-22):2782-90. doi: 10.1016/s0264-410x(03)00181-6. PMID 12798618
- [Background] Biering-Sorensen S, Aaby P, Lund N, Monteiro I, Jensen KJ, Eriksen HB, Schaltz-Buchholzer F, Jorgensen ASP, Rodrigues A, Fisker AB, Benn CS. Early BCG-Denmark and Neonatal Mortality Among Infants Weighing <2500 g: A Randomized Controlled Trial. Clin Infect Dis. 2017 Oct 1;65(7):1183-1190. doi: 10.1093/cid/cix525. PMID 29579158
- [Background] Biering-Sorensen S, Aaby P, Napirna BM, Roth A, Ravn H, Rodrigues A, Whittle H, Benn CS. Small randomized trial among low-birth-weight children receiving bacillus Calmette-Guerin vaccination at first health center contact. Pediatr Infect Dis J. 2012 Mar;31(3):306-8. doi: 10.1097/INF.0b013e3182458289. PMID 22189537
- [Background] Aaby P, Roth A, Ravn H, Napirna BM, Rodrigues A, Lisse IM, Stensballe L, Diness BR, Lausch KR, Lund N, Biering-Sorensen S, Whittle H, Benn CS. Randomized trial of BCG vaccination at birth to low-birth-weight children: beneficial nonspecific effects in the neonatal period? J Infect Dis. 2011 Jul 15;204(2):245-52. doi: 10.1093/infdis/jir240. PMID 21673035
- [Background] Schaltz-Buchholzer F, Biering-Sorensen S, Lund N, Monteiro I, Umbasse P, Fisker AB, Andersen A, Rodrigues A, Aaby P, Benn CS. Early BCG Vaccination, Hospitalizations, and Hospital Deaths: Analysis of a Secondary Outcome in 3 Randomized Trials from Guinea-Bissau. J Infect Dis. 2019 Jan 29;219(4):624-632. doi: 10.1093/infdis/jiy544. PMID 30239767
- [Background] Benn CS, Netea MG, Selin LK, Aaby P. A small jab - a big effect: nonspecific immunomodulation by vaccines. Trends Immunol. 2013 Sep;34(9):431-9. doi: 10.1016/j.it.2013.04.004. Epub 2013 May 14. PMID 23680130
- [Background] Kleinnijenhuis J, Quintin J, Preijers F, Joosten LA, Ifrim DC, Saeed S, Jacobs C, van Loenhout J, de Jong D, Stunnenberg HG, Xavier RJ, van der Meer JW, van Crevel R, Netea MG. Bacille Calmette-Guerin induces NOD2-dependent nonspecific protection from reinfection via epigenetic reprogramming of monocytes. Proc Natl Acad Sci U S A. 2012 Oct 23;109(43):17537-42. doi: 10.1073/pnas.1202870109. Epub 2012 Sep 17. PMID 22988082
- [Background] Kleinnijenhuis J, Quintin J, Preijers F, Benn CS, Joosten LA, Jacobs C, van Loenhout J, Xavier RJ, Aaby P, van der Meer JW, van Crevel R, Netea MG. Long-lasting effects of BCG vaccination on both heterologous Th1/Th17 responses and innate trained immunity. J Innate Immun. 2014;6(2):152-8. doi: 10.1159/000355628. Epub 2013 Oct 30. PMID 24192057
- [Background] Higgins JP, Soares-Weiser K, Lopez-Lopez JA, Kakourou A, Chaplin K, Christensen H, Martin NK, Sterne JA, Reingold AL. Association of BCG, DTP, and measles containing vaccines with childhood mortality: systematic review. BMJ. 2016 Oct 13;355:i5170. doi: 10.1136/bmj.i5170. PMID 27737834
- [Background] Roth A, Gustafson P, Nhaga A, Djana Q, Poulsen A, Garly ML, Jensen H, Sodemann M, Rodriques A, Aaby P. BCG vaccination scar associated with better childhood survival in Guinea-Bissau. Int J Epidemiol. 2005 Jun;34(3):540-7. doi: 10.1093/ije/dyh392. Epub 2005 Jan 19. PMID 15659474
- [Background] Berendsen MLT, Oland CB, Bles P, Jensen AKG, Kofoed PE, Whittle H, de Bree LCJ, Netea MG, Martins C, Benn CS, Aaby P. Maternal Priming: Bacillus Calmette-Guerin (BCG) Vaccine Scarring in Mothers Enhances the Survival of Their Child With a BCG Vaccine Scar. J Pediatric Infect Dis Soc. 2020 Apr 30;9(2):166-172. doi: 10.1093/jpids/piy142. PMID 30715451
- [Background] Storgaard L, Rodrigues A, Martins C, Nielsen BU, Ravn H, Benn CS, Aaby P, Fisker AB. Development of BCG Scar and Subsequent Morbidity and Mortality in Rural Guinea-Bissau. Clin Infect Dis. 2015 Sep 15;61(6):950-9. doi: 10.1093/cid/civ452. Epub 2015 Jun 9. PMID 26060293
- [Background] Schaltz-Buchholzer F, Bjerregaard-Andersen M, Oland CB, Golding C, Stjernholm EB, Monteiro I, Aaby P, Benn CS. Early Vaccination With Bacille Calmette-Guerin-Denmark or BCG-Japan Versus BCG-Russia to Healthy Newborns in Guinea-Bissau: A Randomized Controlled Trial. Clin Infect Dis. 2020 Nov 5;71(8):1883-1893. doi: 10.1093/cid/ciz1080. PMID 31677386
- [Background] Stensballe LG, Sorup S, Aaby P, Benn CS, Greisen G, Jeppesen DL, Birk NM, Kjaergaard J, Nissen TN, Pihl GT, Thostesen LM, Kofoed PE, Pryds O, Ravn H. BCG vaccination at birth and early childhood hospitalisation: a randomised clinical multicentre trial. Arch Dis Child. 2017 Mar;102(3):224-231. doi: 10.1136/archdischild-2016-310760. Epub 2016 Jul 21. PMID 27443836
- [Background] Aaby P, Martins CL, Garly ML, Andersen A, Fisker AB, Claesson MH, Ravn H, Rodrigues A, Whittle HC, Benn CS. Measles vaccination in the presence or absence of maternal measles antibody: impact on child survival. Clin Infect Dis. 2014 Aug 15;59(4):484-92. doi: 10.1093/cid/ciu354. Epub 2014 May 14. PMID 24829213
- [Background] Mawa PA, Webb EL, Filali-Mouhim A, Nkurunungi G, Sekaly RP, Lule SA, Prentice S, Nash S, Dockrell HM, Elliott AM, Cose S. Maternal BCG scar is associated with increased infant proinflammatory immune responses. Vaccine. 2017 Jan 5;35(2):273-282. doi: 10.1016/j.vaccine.2016.11.079. Epub 2016 Nov 30. PMID 27914741
- [Background] Lule SA, Mawa PA, Nkurunungi G, Nampijja M, Kizito D, Akello F, Muhangi L, Elliott AM, Webb EL. Factors associated with tuberculosis infection, and with anti-mycobacterial immune responses, among five year olds BCG-immunised at birth in Entebbe, Uganda. Vaccine. 2015 Feb 4;33(6):796-804. doi: 10.1016/j.vaccine.2014.12.015. Epub 2014 Dec 19. PMID 25529292
- [Background] Behr MA. Comparative genomics of BCG vaccines. Tuberculosis (Edinb). 2001;81(1-2):165-8. doi: 10.1054/tube.2000.0253. PMID 11463238
- [Background] Ritz N, Curtis N. Mapping the global use of different BCG vaccine strains. Tuberculosis (Edinb). 2009 Jul;89(4):248-51. doi: 10.1016/j.tube.2009.03.002. Epub 2009 Jun 18. PMID 19540166
- [Background] Ritz N, Dutta B, Donath S, Casalaz D, Connell TG, Tebruegge M, Robins-Browne R, Hanekom WA, Britton WJ, Curtis N. The influence of bacille Calmette-Guerin vaccine strain on the immune response against tuberculosis: a randomized trial. Am J Respir Crit Care Med. 2012 Jan 15;185(2):213-22. doi: 10.1164/rccm.201104-0714OC. Epub 2011 Nov 3. PMID 22071384
- [Background] Anderson EJ, Webb EL, Mawa PA, Kizza M, Lyadda N, Nampijja M, Elliott AM. The influence of BCG vaccine strain on mycobacteria-specific and non-specific immune responses in a prospective cohort of infants in Uganda. Vaccine. 2012 Mar 9;30(12):2083-9. doi: 10.1016/j.vaccine.2012.01.053. Epub 2012 Jan 31. PMID 22300718
- [Background] Favorov M, Ali M, Tursunbayeva A, Aitmagambetova I, Kilgore P, Ismailov S, Chorba T. Comparative tuberculosis (TB) prevention effectiveness in children of Bacillus Calmette-Guerin (BCG) vaccines from different sources, Kazakhstan. PLoS One. 2012;7(3):e32567. doi: 10.1371/journal.pone.0032567. Epub 2012 Mar 9. PMID 22427854
- [Background] Angelidou A, Conti MG, Diray-Arce J, Benn CS, Shann F, Netea MG, Liu M, Potluri LP, Sanchez-Schmitz G, Husson R, Ozonoff A, Kampmann B, van Haren SD, Levy O. Licensed Bacille Calmette-Guerin (BCG) formulations differ markedly in bacterial viability, RNA content and innate immune activation. Vaccine. 2020 Feb 24;38(9):2229-2240. doi: 10.1016/j.vaccine.2019.11.060. Epub 2020 Jan 28. PMID 32005538
- [Background] Veirum JE, Sodeman M, Biai S, Hedegard K, Aaby P. Increased mortality in the year following discharge from a paediatric ward in Bissau, Guinea-Bissau. Acta Paediatr. 2007 Dec;96(12):1832-8. doi: 10.1111/j.1651-2227.2007.00562.x. PMID 18001338
- [Background] Biai S, Rodrigues A, Nielsen J, Sodemann M, Aaby P. Vaccination status and sequence of vaccinations as risk factors for hospitalisation among outpatients in a high mortality country. Vaccine. 2011 May 9;29(20):3662-9. doi: 10.1016/j.vaccine.2011.03.016. Epub 2011 Apr 6. PMID 21440640
- [Background] Bamji M, Stone RK, Kaul A, Usmani G, Schachter FF, Wasserman E. Palpable lymph nodes in healthy newborns and infants. Pediatrics. 1986 Oct;78(4):573-5. PMID 3763263
- [Background] Roloff V, Higgins JP, Sutton AJ. Planning future studies based on the conditional power of a meta-analysis. Stat Med. 2013 Jan 15;32(1):11-24. doi: 10.1002/sim.5524. Epub 2012 Jul 11. PMID 22786670
- [Background] Stefanova T. Quality control and safety assessment of BCG vaccines in the post-genomic era. Biotechnol Biotechnol Equip. 2014 May 4;28(3):387-391. doi: 10.1080/13102818.2014.927200. Epub 2014 Jul 10. PMID 26019525
- [Background] Wada T, Maruyama F, Iwamoto T, Maeda S, Yamamoto T, Nakagawa I, Yamamoto S, Ohara N. Deep sequencing analysis of the heterogeneity of seed and commercial lots of the bacillus Calmette-Guerin (BCG) tuberculosis vaccine substrain Tokyo-172. Sci Rep. 2015 Dec 4;5:17827. doi: 10.1038/srep17827. PMID 26635118
- [Background] Bottai D, Brosch R. The BCG Strain Pool: Diversity Matters. Mol Ther. 2016 Feb;24(2):201-203. doi: 10.1038/mt.2016.18. No abstract available. PMID 26906614
- [Background] Ritz N, Hanekom WA, Robins-Browne R, Britton WJ, Curtis N. Influence of BCG vaccine strain on the immune response and protection against tuberculosis. FEMS Microbiol Rev. 2008 Aug;32(5):821-41. doi: 10.1111/j.1574-6976.2008.00118.x. Epub 2008 Jul 9. PMID 18616602
- See also: WHO data regarding child mortality. — http://www.who.int/gho/child_health/mortality/neonatal_text/en/
- See also: The BCGSTRAIN II trial from which the results have not yet been published (follow-up is still pending and will be finished by october 2020). — https://clinicaltrials.gov/ct2/show/NCT03400878
- See also: Description of the verbal autopsy instrument which will be used for HDSS infants included in the trial. — https://cdn.who.int/media/docs/default-source/mca-documents/verbal-autopsy-standards-the-2012-who-verbal-autopsy-instrument---release-candidate-1.pdf?sfvrsn=68f9b5a4_1&download=true
- See also: Evidence based recommendations on non-specific effects of BCG, DTP-containing and measles-containing vaccines on mortality in children under 5 years of age. Background paper for SAGE discussions — https://terrance.who.int/mediacentre/data/sage/SAGE_Docs_Ppt_Apr2014/9_session_non-specific_vaccine_effects/Apr2014_session9_non-specific_vaccine_effects.pdf